CLINICAL TRIAL: NCT04111146
Title: The Clinical Effect of Preoperative Level of 25-OH-vitamin D3 on the Liver Transplant Recipients
Brief Title: Effect of 25-OH-vitamin D3 on the Liver Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyung, Professor, Asan Medical Center
Other Study IDs: AsanMC-vitamin D
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Liver Transplant Disorder
Keywords: vitamin D; liver transplant; hospital stay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Liver transplant patients with severe vitamin D deficiency (<10ng/ml)
- 2: Liver transplant patients with vitamin D insufficiency (10-20ng/ml)
- 3: Liver transplant patients with normal vitamin D status (>20ng/ml)

SUMMARY:
The low vitamin D3 levels and malnutrition before liver transplantation showed an increase in the length of stay in ICU and hospital. Although several factors may influence the clinical outcomes of patients with liver transplantation, low vitamin D3 levels showed an independent risk factor. It is necessary to prospectively analyze the effect of vitamin D supplements on clinical outcomes in liver transplant recipients.

DETAILED DESCRIPTION:
Purpose: Vitamin D deficiency is common in patients of chronic liver disease and has been associated with infection and mortality. The aim of this study is to determine whether preoperative vitamin D levels affect clinical outcomes after liver transplantation.

Methods : This was a single-center retrospective study. Between June and November 2017, a total of 219 patients underwent liver transplantation. The primary outcome was the relationship between serum 25-OH-vitamin D3 level before liver transplantation and length of stay in the intensive care unit (ICU). Secondary outcomes included the duration of normalization of inflammatory marker, such as white blood cell count (WBC) & C-reactive protein (CRP) after liver transplantation, new infection rates, rejection rates, the length of hospital stay and mortality among vitamin D level.

ELIGIBILITY:
Inclusion Criteria:

* The patients who admitted to intensive care unit (ICU) after liver transplantation were studied

Exclusion Criteria:

* Patients who didn't have preoperative vitamin D level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients received liver transplantation from June 2017 to November 2017
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Hospital stay after liver transplant | 6 months
  compared with each group

SECONDARY OUTCOMES:
duration of normalization of CRP, WBC | 6 months
  compared with each group
Length of ICU stay | 6 months
  compared with each group
New infection rate | 6 months
  compared with each group

CONTACTS AND LOCATIONS:
Locations (1):
- Hakjae Lee, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finkelmeier F, Kronenberger B, Koberle V, Bojunga J, Zeuzem S, Trojan J, Piiper A, Waidmann O. Severe 25-hydroxyvitamin D deficiency identifies a poor prognosis in patients with hepatocellular carcinoma - a prospective cohort study. Aliment Pharmacol Ther. 2014 May;39(10):1204-12. doi: 10.1111/apt.12731. Epub 2014 Mar 29. PMID 24684435
- [Result] Finkelmeier F, Kronenberger B, Zeuzem S, Piiper A, Waidmann O. Low 25-Hydroxyvitamin D Levels Are Associated with Infections and Mortality in Patients with Cirrhosis. PLoS One. 2015 Jun 29;10(6):e0132119. doi: 10.1371/journal.pone.0132119. eCollection 2015. PMID 26121590
- [Result] Grant C. A vitamin D protocol post-liver transplantation. J Am Assoc Nurse Pract. 2017 Nov;29(11):658-666. doi: 10.1002/2327-6924.12503. Epub 2017 Aug 25. PMID 28840965
- [Result] Zhou Q, Li L, Chen Y, Zhang J, Zhong L, Peng Z, Xing T. Vitamin D supplementation could reduce the risk of acute cellular rejection and infection in vitamin D deficient liver allograft recipients. Int Immunopharmacol. 2019 Oct;75:105811. doi: 10.1016/j.intimp.2019.105811. Epub 2019 Aug 15. PMID 31422183